CLINICAL TRIAL: NCT03756389
Title: An Exploratory Trial to Evaluate the Clinical Effectiveness of a Topical Application of BMX-010 in Subjects With Rosacea
Brief Title: Evaluation of Topical Application of BMX-010 in Subjects With Rosacea
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Re-formulation of study product
Sponsor: BioMimetix JV, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMX-DERM-202
Record Dates: First submitted 2018-11-15; First posted 2018-11-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Masking Description: In Part A, all subjects will receive study drug and this is Open Label. When Part A is complete, Part B will start and this will be double blind to participant and investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMX-010 0.03% (Experimental): Approximately 30 subjects will receive BMX-010 0.03% for 7-28 days to be applied topically to Rosacea of the face.
  Interventions: Drug: BMX-010
- BMX-010 0.1% (Experimental): Approximately 30 subjects will receive BMX-010 0.1% for 7-28 days to be applied topically to Rosacea of the face.
  Interventions: Drug: BMX-010

INTERVENTIONS:
Drug: BMX-010 — Safety and efficacy of BMX-010 in topical treatment of rosacea.

SUMMARY:
This is an exploratory Phase 2 trial of BMX-010 in patients with Rosacea which will be conducted in two parts. Up to 210 subjects with Rosacea will be enrolled.

DETAILED DESCRIPTION:
Part A is designed to confirm the optimal formulation, strength, and dosing frequency of the study drug. Up to 60 subjects will be enrolled in this part.

Part B is designed to be a randomized, double-blind trial studying the optimal formulation, strength, and dosing frequency of BMX-010 as determined in Part A, compared to Placebo. Up to 150 subjects will be enrolled in this part.

In both parts, adult subjects with Rosacea will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age;
2. A clinical diagnosis of mild to severe facial rosacea;
3. Screening and Baseline IGA score > 2 (greater than or equal to 2);
4. A minimum Clinician Erythema Assessment (CEA) score of 2 at Screening and at Baseline Visits (prior to the investigational product application);
5. Willing to refrain from using any topical or systemic treatments for inflammatory skin disease, other than the investigational product;
6. Candidate for topical treatment of Rosacea;
7. If a cleanser, moisturizer or sunscreen is needed during the study, Subjects must be willing to use only allowed cleansers, moisturizers, sunscreens, or moisturizer/sunscreen combination products. If the subject wears makeup they must agree to use non-comedogenic makeup;
8. Females of child-bearing potential must have a negative urine pregnancy test within 48 hours prior to the first drug administration;
9. Females of child-bearing potential must be willing to use 2 methods of contraception deemed adequate by the investigator (for example, oral contraceptive pills plus a barrier method) through the trial and for 1 month thereafter to be eligible for, and continue participation in, the study;
10. Ability to complete the study in compliance with the protocol, including agreement in writing to apply study product only to the assigned areas; and
11. Ability to understand and provide written informed consent.

Exclusion Criteria:

1. Any dermatological conditions on the face that could interfere with clinical evaluations;
2. Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive;
3. Presence of beard or excessive facial hair at Screening which would interfere with the study treatments or study assessments and refusal to remove for duration of study;
4. Subjects with any underlying disease that the Investigator deems uncontrolled, and poses a concern for the subject's safety while participating in the study;
5. Concomitant skin disease that could confound clinical evaluations or increase risk to the subject;
6. Use of medicated make-up (including anti-aging make-up) throughout the study;
7. Use during the study of 1) systemic steroids, 2) topical retinoids to the face, 3) antibiotics known to impact rosacea, 4) immunosuppressive agents, or immunomodulators;
8. Facial use of 1) topical steroids, 2) topical anti-inflammatory agents, 3) topical antimycotics, 4) any topical rosacea treatments or 4) topical antibiotics;
9. Use of medicated cleansers on the face (throughout the study);
10. Use of topical astringents or abrasives, medical topical preparations (prescription and OTC products) within 2 days prior to Baseline and throughout the study;
11. Systemic or skin infection requiring antimicrobial therapy;
12. Systemic chemotherapy or radiotherapy within 4 weeks of the Baseline Visit;
13. Immunocompromise of any cause, known human immunodeficiency virus infection, or acquired immunodeficiency syndrome;
14. Pregnancy, planned pregnancy, lactation, or inadequate contraception as judged by the investigator;
15. Active drug or alcohol dependence;
16. Significant acute or chronic medical, neurological, or psychiatric illness that, in the judgment of the investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study;
17. Previous clinical trial participation for the indication being treated in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-03 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Determine whether the optimum frequency of topical application of BMX-010 0.03% is once per day or twice per day for a treatment interval of up to 28 days. | 28 days
  Assessed by number of participants with a change in Investigator Global Assessment (IGA) grade which will be assessed weekly.
Determine whether the optimum frequency of topical application of BMX-010 0.03% is once per day or twice per day for a treatment interval of up to 28 days. | 28 days
  Assessed by number of participants with a change in Clinical Erythema Assessment (CEA) grade which will be assessed weekly.
Determine whether the optimum frequency of topical application of BMX-010 0.1% is once per day or twice per day for a treatment interval of up to 28 days. | 28 days
  Assessed by number of participants with a change in Investigator Global Assessment (IGA) grade which will be assessed weekly.
Determine whether the optimum frequency of topical application of BMX-010 0.1% is once per day or twice per day for a treatment interval of up to 28 days. | 28 days
  Assessed by number of participants with a change in Clinical Erythema Assessment (CEA) grade which will be assessed weekly.
Determine if BMX-010 cream or gel provides better efficacy in the treatment of rosacea. | 43 days
  Assessed by number of participants with a change in Investigator Global Assessment (IGA) grade. This will be assessed weekly with a final assessment two weeks after dosing ends (Day 43).
Determine if BMX-010 cream or gel provides better efficacy in the treatment of the redness of rosacea. | 43 days
  Assessed by number of participants with a change in Clinical Erythema Assessment (CEA) grade. This will be assessed weekly with a final assessment two weeks after dosing ends (Day 43).
Evaluate the efficacy of BMX-010 in treatment of rosacea. | 43 days
  Assessed by number of participants with a change in Investigator Global Assessment (IGA) grade. This will be assessed weekly with a final assessment two weeks after dosing ends (Day 43).
Evaluate the effect of BMX-010 on redness in patients with rosacea. | 43 days
  Assessed by number of participants with a change in Clinical Erythema Assessment (CEA) grade. This will be assessed weekly with a final assessment two weeks after dosing ends (Day 43).

SECONDARY OUTCOMES:
Document, as possible, the clinical effects of BMX-010 in subjects with Rosacea through clinical photography. | 43 days
  If consented by the patient, photos will be taken at each study visit.
Assess the mean percent reduction change in inflammatory papules/pustules counts from baseline to end of study. | 43 days
  Inflammatory lesions will be counted at each study visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado Skin Care, Englewood, Colorado, United States